CLINICAL TRIAL: NCT01501695
Title: A 3-arm Phase III Study of 5LGr, Tiapride or Placebo in Pediatric Patients With Tic Disorder
Brief Title: Phase III Study of 5LGr to Treat Tic Disorder
Acronym: 5LGr
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCT00797953
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Tic Disorder; Tourette Syndrome; Chronic Tic Disorder
Keywords: tic disorder; pediatric
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome | interventions — Tiapride Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5LGr, granule and placebo tablet (Experimental): Drug:5LGr; Dosage form:Granule;Strength:5 gram/sack;Mimic Tablet:0 mg/tablet. Dosage: 5LGr Granule: 1 sack, t.i.d. for patients less than 12 yrs,whereas 1.5 sacks, t.i.d. for patients 13-18 yrs.
  Mimic tablet:For patients 5-12 yrs: 0.5 tablet, b.i.d for first 2 weeks, then 1 tablet, bid for next 6 weeks; for patients 13-18 yrs: tablet b.i.d for first 2 weeks, then 2 tablets b.i.d for next 6 weeks.
  Duration: 8 weeks.
  Interventions: Drug: 5LGr
- tiapride tabletand mimic 5LGr granule (Active Comparator): Tiapride are 100 mg scored tablets. Mimic 5LGr granule are preparation that contain no active ingredient, and act as placebo.
  Dosage: Tiaptride tablet: For patients 5-12 yrs: 50mg bid for first 2 weeks, then 100 mg, bid for next 6 weeks; for patients 13-18 yrs:100mg bid for first 2 weeks, then 200 mg bid for next 6 weeks.
  Mimic 5LGr Granule:Strength:0 gram/sack.Dosage:1 sack for patients less than 12 yrs,while 1.5 sacks for patients 13-18 yrs.Frequency: T.i.d.
  Duration: 8 weeks.
  Interventions: Drug: tiapride
- placebo, granule and tablet (Placebo Comparator): This arm includes mimic preparation of 5LGr granule and tiapride tablets , which doesn't contain active ingredients.
  Dosage form: Mimic Granule:Strength:0 gram/sack Dosage:1 sack, t.i.d for patients less than 12 yrs,while 1.5 sacks, t.i.d for patients 13-18 yrs.
  Mimic tablet:Strength:0 mg/tablet.For patients 5-12 yrs: 0.5 tablets b.i.d for first 2 weeks, then 1 tablet,b.i.d for next 6 weeks; for patients 13-18 yrs:1 tablet b.i.d for first 2 weeks, then 2 tablets b.i.d for next 6 weeks.
  Duration: 8 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 5LGr — Dosage form:Granule Strength:5 gram/sack Dosage:1 sack for patients less than 12 yrs 1.5 sacks for patients 13-18 yrs. Frequency: three times per day. Duration: 8 weeks.
  Other Names: Wuling Granule
  Arms: 5LGr, granule and placebo tablet
Drug: tiapride — dosage form: tablet Strength:100 mg Dosage: For patients 5-12 yrs: 50mg bid for first 2 weeks, then 100 mg, bid for next 6 weeks; for patients 13-18 yrs:100mg bid for first 2 weeks, then 200 mg bid for next 6 weeks.
  Total duration:8 weeks.
  Other Names: Tiapridel, Tiapridax
  Arms: tiapride tabletand mimic 5LGr granule
Drug: placebo — mimetic granule: same with 5LGr mimetic tablet: same with tiapride
  Other Names: Blank tablet
  Arms: placebo, granule and tablet

SUMMARY:
The purpose of this study is to evaluate the effective and safety of 5LGr in pediatric patients with tic disorders.

DETAILED DESCRIPTION:
5LGr is a kind of traditional Chinese medicine(TCM) which under the direction of TCM theory.The aim of this study is prove the effective and safety of 5LGr in children and adolescence of Tic syndrome sub-population with specific TCM syndrome differentiation, when compared with tiapride and placebo.

ELIGIBILITY:
Inclusion Criteria:

* >1 year history of diagnosed tic disorder;
* age:5-18 yrs;
* YGTSS score>=30 at baseline.

Exclusion Criteria:

* Diagnosed with hyperactivity disorder,epilepsy,chorea,autism,obsessive-compulsive disorder,mental retardation,athetosis,Wilson's disease.
* Any indefinite tic disorder or tic disorders caused by medication.
* Participation to other studies.
* Patients with loose stool.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 603 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale(YGTSS) score change from baseline at 8 weeks | Within 8 weeks of completion intervention.
  The outcome will be assessed at 8th weeks. And patients who judged as effective by investigator will be included in a follow-up period up to 4 weeks.

SECONDARY OUTCOMES:
Change of syndrome scales from baseline at 8 weeks; | Within 8 weeks of completion intervention.
Change of YGTSS scores from baseline at 2 weeks; | within 2 weeks of intervention
Change of syndrome scales from baseline at 2 weeks; | Within 2 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Xinmin Han, M.D., Principal Investigator — Nanjing University of TCM affiliated hospital; Yi zheng, Principal Investigator — Capital Medical University; Minjie Wang, M.D., Principal Investigator — Nanjing Medical college Attached Brain Branch Hospital; Xiaowei Wei, M.D., Principal Investigator — First Teaching Hospital of Tianjin University of Traditional Chinese Medicine; Yan Cheng, M.D., Principal Investigator — Second Teaching Hospital of Tianjin University of Traditional Chinese Medicine; Xuefeng Wang, M.D., Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; Yuyan Chen, M.D., Principal Investigator — Zhejiang University of TCM affiliated hospital; Ying Ding, M.D., Principal Investigator — Henan University of TCM affiliated hospital

REFERENCES:
- [Derived] Zheng Y, Zhang ZJ, Han XM, Ding Y, Chen YY, Wang XF, Wei XW, Wang MJ, Cheng Y, Nie ZH, Zhao M, Zheng XX. A proprietary herbal medicine (5-Ling Granule) for Tourette syndrome: a randomized controlled trial. J Child Psychol Psychiatry. 2016 Jan;57(1):74-83. doi: 10.1111/jcpp.12432. Epub 2015 Jun 13. PMID 26072932
- See also: Manufacturer — http://www.tasly.com